CLINICAL TRIAL: NCT05806827
Title: CONNECTED - INVESTIGATE THE ASSOCIATION BETWEEN VIRAL NEUROTOXIC INFECTION AND POSTOPERATIVE DELIRIUM AND POSTOPERATIVE COGNITIVE DECLINE
Brief Title: INVESTIGATE THE ASSOCIATION BETWEEN VIRAL NEUROTOXIC INFECTION AND POSTOPERATIVE DELIRIUM AND POSTOPERATIVE COGNITIVE DECLINE
Acronym: CONNECTED
Status: Not yet recruiting | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Federico Bilotta, Professor, University of Roma La Sapienza
Other Study IDs: CONNECTED-ObsCT
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: POSTOPERATIVE DELIRIUM AND POSTOPERATIVE COGNITIVE DECLINE

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collection of peripheral blood and serum specimen
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Virological screening — The preoperative viral screening protocol will start with a self-assessment questionnaire that will be provided to all the enrolled patients, where they will be asked to indicate previously SARS-CoV-2, HPV, EBV, CMV infections. Collection of peripheral blood mononuclear cells (PBMCs) from blood samples and serum specimens for the virological screening (HPV, EBV, CMV, SARS-CoV-2). Preoperative MoCA assessment, follow-up 5 days, 3 months and 6 months after the surgery.
  Other Names: cognitive assessment

SUMMARY:
In the last two decades, viral infections have increased dramatically : the 2003 severe acute respiratory syndrome coronavirus outbreak, the 2009 swine flu pandemic, the 2012 Middle East respiratory syndrome coronavirus outbreak, the 2013-2016 Ebola virus disease epidemic in West Africa and the 2015 Zika virus disease epidemic and not least the COVID-19 pandemic.

At the same time, neurological disorders are a major and increasing global health challenge, which accounts for a substantial portion of the disease burden worldwide . In Europe, more than half of the population (approx. 60% ) suffers from a neurological disease, ranking number three among all disease groups . The figures are higher in the population with more than 65 years.

Based on Eurostat annual publication "Aging Europe", in 2020 people over 65 represented 20.6% of the European Union population, and the projections show that the share of people over 65 is expected to strongly increase until 2058, reaching 30.3% of the EU population.

Furthermore, while in civil aviation, the mortality rate is estimated around 0,00525% (Eurocontrol, 2022), the perioperative mortality rate in Europe is about 4% (Pearse et al., 2012). Clearly, the patients undergoing surgery already have a higher mortality risk depending on their initial medical conditions. However, the medical field can without doubts benefit from an improved risks assessment approach derived from the civil aviation.

Against this backdrop, the project aims at:

i) researching the correlation between a neurotoxic viruses' infection and the increased risk, in terms of frequency or severity, of developing a cognitive disfunction such as the postoperative cognitive dysfunction (POCD), by conducting an observational clinical trial on selected neurotoxic viruses (SARS-CoV-2, Herpes simplex virus, Cytomegalovirus and Epstein Barr virus).

ii) developing a theoretical model for monitoring the implications of general anaesthesia in elder patients aged ≥ 65 years iii) designing a risk assessment mechanism, based on the best practices developed in the aerospace sector, for patients with neurotoxic infection and POCD, that can be furtherly scalable in other medical contexts.

iv) building an AI-based platform, following the example of the NSQIP risk calculator for cardiovascular postoperative complications, both for data collection and data processing, able to return an estimate of the risk of perioperative-related cognitive complications in elder patients undergoing major elective surgeries.

Observational Clinical Trial The clinical trial will recruit a sample of 1685 patients in eight centres (about 250 patients per centre, considering also the drop-out rate) to be finalised in 24 months.

The primary end point of the clinical trial is to evaluate if patients undergoing general anaesthesia for elective major surgeries lasting longer than 1 hour that have an history of COVID-19 (not an active SARS-CoV-2 infection) do have a higher risk to develop postoperative cognitive dysfunction (POCD)/delayed neurocognitive recovery (DNC) at 3 months and 6 months follow up after surgery.

Secondary end point include:

1. - Relationship between POCD/DNC with preoperative exposure to other neurotropic viruses: Herpes simplex virus (HS), Cytomegalovirus (CMV), and Epstein Barr virus (EBV).
2. - Development -on the basis of collected data- of a software dedicated to calculating in the preoperative phase the risk for early postoperative delirium or POCD/PNDs.
3. - Development of a conceptual model of "perioperative safety management": as in civil aviation traffic control, increasing the patients' perception of healthcare safety and quality.
4. - Delivery of training to healthcare practitioners concerning the preoperative evaluation of POD risk and the identification of patients at risk.

ELIGIBILITY:
The recruitment's inclusion criteria will select patients:

* Aged ≥ 65 years
* Undergoing elective surgical procedures, scheduled to last longer than one hour.
* Under general anaesthesia, including the procedures using mechanical ventilation, total intravenous anaesthesia (TIVA) or balanced anaesthesia.
* Planned inpatient length of stay in the hospital ≥ 2 days
* With and without preoperative exposure to the following neurotoxic viruses: SARS-CoV-2 (COVID-19), Herpes simplex virus (HS), Cytomegalovirus (CMV), and Epstein Barr virus (EBV).

Exclusion Criteria:

* Patients aged less than 65 years old.
* Undergoing non elective surgical procedures.
* Undergoing surgical procedures lasting less than one hour.
* Undergoing surgical procedures entailing the impairment of the verbal production, such as brain surgery, maxillofacial surgery and otorhinolaryngology operations. The surgical procedures excluded are the ones affecting the speech and cognitive functions and the surgeries with specific risks of postoperative cognitive impairment (such as cardiac surgery and carotid surgery).
* Undergoing surgical procedures implying local anaesthesia.
* Undergoing surgical procedures that do not imply the insertion of an airway device (such as endotracheal tube or laryngeal mask) or the protracted mechanical ventilation.
* Undergoing surgery procedures with planned mechanical ventilation after surgery / re-intubation.
* Patients with language barriers.
* Patients under legal guardianship and with pre-existing cognitive dysfunction (MoCA < 21 points).
* Patients not giving the informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: candidates aged ≥ 65 years underging major elective surgery under general anaesthesia
Sampling Method: Probability Sample
Enrollment: 1685 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
ASSOCIATION BETWEEN VIRAL NEUROTOXIC INFECTION AND POSTOPERATIVE DELIRIUM AND POSTOPERATIVE COGNITIVE DECLINE | 24 months
  to evaluate if patients undergoing general anaesthesia for elective major surgeries lasting longer than 1 hour that have an history of COVID-19 (not an active SARS-CoV-2 infection) do have a higher risk to develop postoperative cognitive dysfunction (POCD)/delayed neurocognitive recovery (DNC) at 3 months and 6 months follow-up after surgery.

SECONDARY OUTCOMES:
Association between POCD/DNC and HSV/CMV/EBV | 24 months
  Association between POCD/DNC with preoperative exposure to other neurotropic viruses: Herpes simplex virus (HS), Cytomegalovirus (CMV), and Epstein Barr virus (EBV).
POCD risk calculator | 24 months
  Development -on the basis of collected data- of a software dedicated to calculating in the preoperative phase the risk for early postoperative delirium or POCD/PNDs
perioperative safety management | 24 months
  Development of a conceptual model of "perioperative safety management": as in civil aviation traffic control, increasing the patients' perception of healthcare safety and quality.
training of healthcare practitioners | 24 months
  Delivery of training to healthcare practitioners concerning the preoperative evaluation of POD risk and the identification of patients at risk.

IPD SHARING:
Plan to Share IPD: Undecided